CLINICAL TRIAL: NCT05526300
Title: Randomized Study of Antihypertensive Intervention by Intelligent Hypertension Management System
Brief Title: Intelligent Hypertension Intervention Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Tong Ren Hospital (Other)
Responsible Party: Principal Investigator, Hou Lei, Director of cardiovascular disease institute, Shanghai Tong Ren Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ShanghaiTRH-hypertension
Record Dates: First submitted 2022-08-31; First posted 2022-09-02 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2024-12

CONDITIONS: To Explore Whether the Application of Intelligent Hypertension Management System Can Effectively Reduce Blood Pressure in Hypertensive Patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The standard care group (Active Comparator)
  Interventions: Other: The standard care
- Intelligent intervention group (Experimental)
  Interventions: Device: Intelligent Hypertension Management System

INTERVENTIONS:
Device: Intelligent Hypertension Management System — The intelligent hypertension management system is used to remotely detect the blood pressure of hypertensive patients
  Arms: Intelligent intervention group
Other: The standard care — The standard care
  Arms: The standard care group

SUMMARY:
To explore whether the application of intelligent hypertension management system can effectively reduce blood pressure in hypertensive patients. A total of 320 eligible subjects will be recruited and randomization to two groups. The standard care group (n=160) will receive conventional hypertension treatment with baseline data collected.Wearable blood pressure monitoring device management group (intervention group, n=160) will receive blood pressure monitoring remotely everyday and antihypertension medication treatment. Primary outcome is Net change in systolic blood pressure from baseline to 3 months follow-up. Secondary outcomes include Net change in diastolic blood pressure hypertension control ratio (BP < 140/90 mmHg)

ELIGIBILITY:
Inclusion Criteria:

1. Aged more than 18 years old, less than or equal to 75 years old.
2. Hypertensive patients (systolic/diastolic blood pressure ≥140/90 mmHg at two separate screening/baseline visits)
3. Patients or guardians can skillfully use devices such as smartphones and electronic sphygmomanometers
4. Voluntarily joined and signed the informed consent

Exclusion Criteria:

1. Pregnant women or women planning to become pregnant within the next year;
2. Patients with secondary hypertension
3. Patients with life expectancy less than 1 year
4. Severe hepatic and renal insufficiency (ALT > 5 times ULA, eGFR < 15ml/min/1.73mm2)
5. Known active malignancy disease
6. The researcher believes that patients who are not suitable to participate in this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2022-09-06 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Net change in systolic blood pressure from baseline to 3 months follow-up | one and three months after study

SECONDARY OUTCOMES:
Net change in diastolic blood pressure | one and three months after study
Hypertension control ratio (BP < 140/90 mmHg) | one and three months after study

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Shanghai tongren hospital, Shanghai, Shanghai Municipality
  - Shanghai Fifth Rehabilitation Hospital, Shanghai
  - Songjiang hospital, Shanghai jiaotong University, School of medicine, Shanghai

IPD SHARING:
Plan to Share IPD: Yes
The data that support the findings of this study are available in ClinicalTrials. gov at https://register.clinicaltrials.gov/prs/app/action/SelectProtocol?sid=S000CFXV&selectaction=Edit&uid=U0004XRB&ts=32&cx=-oc8exc. And can be accessed with reference number: NCT05526300. The individual deidentified participant data (including data dictionaries) will be available. All of the individual participant data collected during the trial will be shared after de-identification. The study protocol, and statistical analysis plan will be available. The data will become available Immediately following publication and with no end date. The data will be shared with researchers who wish to access the data to help patients for non-profit purposes. Data are available indefinitely at ClinicalTrials. gov.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will become available Immediately following publication and with no end date. T
Access Criteria: The data will be shared with researchers who wish to access the data to help patients for non-profit purposes.

REFERENCES:
- [Derived] Yu H, Chen X, Xia J, Hou L. Effect of intelligent hypertension management system on blood pressure: protocol for a randomised controlled multicentre trial. BMJ Open. 2023 Dec 12;13(12):e074580. doi: 10.1136/bmjopen-2023-074580. PMID 38086588